CLINICAL TRIAL: NCT05626231
Title: Development of a Training Intervention to Improve Mental Health Treatment Effectiveness and Engagement for Youth With Documented Mental Health Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Training Development Study; K23MH124670 (NIH)
Record Dates: First submitted 2022-11-01; First posted 2022-11-23 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: youth; child; adolescent; young adult; psychologist; social worker; psychiatrist; counselor; teen; provider; therapist; clinician
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: The single-arm intervention will test an online, asynchronous training intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training Intervention (Experimental): The single-arm intervention study will test an online asynchronous evidence-based practices training intervention.
  Interventions: Behavioral: Training Intervention

INTERVENTIONS:
Behavioral: Training Intervention — The training intervention is a modular online asynchronous training intervention designed to increase mental health providers' use of evidence-based practices with youth patients (ages 12-25). It was developed using community-engaged and human-centered design methods with key stakeholders (youth, their parents, mental health providers). In this open trial, the training will be offered to mental health providers at a multisite mental health clinic in the U.S. (referred to as "pilot site" herein).

SUMMARY:
The overall goal of the larger 3-aim study is to develop and pilot test a training intervention to increase mental health providers' use of evidence-based practices with youth patients. Aim 3 (registered here) of the study is an open trial pilot study at a multi-clinic mental health agency, aimed at examining the feasibility and acceptability of conducting a future randomized controlled trial (RCT).

DETAILED DESCRIPTION:
The overall goal of the larger 3-aim study is to develop and pilot test a training intervention to increase mental health providers' use of evidence-based practices with youth patients. The Boston College Institutional Review Board (IRB) approved protocol #21.247.01-15. Aim 1 involved designing the training intervention through an extensive literature review and community-engaged methods that centered on collaborations with providers, youth patients, and parents. Aim 2 (in progress) entails refining the training intervention via human centered design methods. Aim 3 (registered here) of the study is an open trial pilot study at a multi-clinic mental health agency, aimed at examining the feasibility and acceptability of conducting a future randomized controlled trial (RCT). Effectiveness and implementation data from both providers (n=49) and patients (i.e., youth and their parents; n=50 GMY and n=30 caregivers) will be collected and analyzed. Primary outcomes are measured at the provider-level and secondary outcomes are measured at the patient-level (i.e., patients and their parents).

ELIGIBILITY:
Inclusion Criteria:

For provider participants:

* Mental health care providers (e.g., psychologists, social workers) employed by the pilot site at the time of the pilot test and who work with clients ages 12-25
* Age 18 or older
* Fluent in English

For GMY participants:

* Identify as a gender-minority.
* Age 12-25
* Currently receiving mental health services from the pilot site
* Fluent in English

For parents of youth participants:

* Parents of youth currently receiving mental health services at the pilot site
* 18 or older
* Fluent in English

Exclusion Criteria:

* Provided that participants meet the aforementioned inclusion criteria, there are no explicit criteria for exclusion.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Youth participants will have gender-based inclusion criteria. The youth must identify as a gender-minority.
Enrollment: 286 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maggi Price, PhD, Principal Investigator — Boston College School of Social Work
Locations (1):
- Boston College, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bidell MP. The Sexual Orientation Counselor Competency Scale: Assessing attitudes, skills, and knowledge of counselors working with lesbian, gay, and bisexual clients. Counselor Education and Supervision. 2011; 44(4): 267-279.
- [Background] Pachankis JE, Soulliard ZA, Seager van Dyk I, Layland EK, Clark KA, Levine DS, Jackson SD. Training in LGBTQ-affirmative cognitive behavioral therapy: A randomized controlled trial across LGBTQ community centers. J Consult Clin Psychol. 2022 Jul;90(7):582-599. doi: 10.1037/ccp0000745. PMID 35901370
- [Background] Athay MM, Bickman L. Development and psychometric evaluation of the youth and caregiver Service Satisfaction Scale. Adm Policy Ment Health. 2012 Mar;39(1-2):71-7. doi: 10.1007/s10488-012-0407-y. PMID 22407558
- [Background] Duppong Hurley K, Lambert MC, Van Ryzin M, Sullivan J, Stevens A. Therapeutic Alliance Between Youth and Staff in Residential Group Care: Psychometrics of the Therapeutic Alliance Quality Scale. Child Youth Serv Rev. 2013 Jan 1;35(1):56-64. doi: 10.1016/j.childyouth.2012.10.009. Epub 2012 Nov 8. PMID 23264715
- [Background] Bickman L, Kelley SD, Breda C, de Andrade AR, Riemer M. Effects of routine feedback to clinicians on mental health outcomes of youths: results of a randomized trial. Psychiatr Serv. 2011 Dec;62(12):1423-9. doi: 10.1176/appi.ps.002052011. PMID 22193788
- [Background] Bickman L, Douglas SR, De Andrade AR, Tomlinson M, Gleacher A, Olin S, Hoagwood K. Implementing a Measurement Feedback System: A Tale of Two Sites. Adm Policy Ment Health. 2016 May;43(3):410-25. doi: 10.1007/s10488-015-0647-8. PMID 25876736
- [Derived] Price MA, Mulkern PJ, Condon M, Rakhilin M, Johansen K, Lyon AR, Saldana L, Pachankis J, Woodward SA, Roeder KM, Moran LR, Jerskey BA. Leveraging community engagement and human-centered design to develop multilevel implementation strategies to enhance adoption of a health equity intervention. Implement Sci Commun. 2025 Nov 24;6(1):130. doi: 10.1186/s43058-025-00809-7. PMID 41287012
- [Derived] Price MA, Mulkern PJ, Condon M, Rakhilin M, Johansen K, Lyon AR, Saldana L, Pachankis J, Woodward SA, Roeder KM, Moran LR, Jerskey BA. Leveraging Community Engagement and Human-Centered Design to Develop Multilevel Implementation Strategies to Enhance Adoption of a Health Equity Intervention. Res Sq [Preprint]. 2025 Mar 28:rs.3.rs-5702080. doi: 10.21203/rs.3.rs-5702080/v1. PMID 40195981

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Providers were not actively recruited, but rather, all partner clinic mental health providers (e.g., psychiatrists, social workers) were invited to participate in the study.
  Youth patients and their parents recruitment involved sending an interest email to the partner clinic's listserv of all patients and paretnss. Otherwise, youth will be included in the study if they received treatment at the clinic during the open trial phase and were between the ages of 12-25.
Groups:
- Training Intervention: The single-arm intervention study will test an online asynchronous evidence-based training intervention called
  The training is a modular online asynchronous training intervention designed to increase mental health providers' use of evidence-based practices with youth patients (ages 12-25). It was developed using community-engaged and human-centered design methods with key stakeholders (youth, their parents, mental health providers). In this open trial, the training will be offered to mental health providers at a multisite mental health clinic in the U.S. (referred to as "pilot site" herein).
Period: Provider Enrollment
Arm/Group | Training Intervention
Started | 109 (Providers at partner clinic identified as eligible for the study)
Providers Who Consented to the Study | 93
Completed | 93
Not Completed | 16
Not completed — Worked part-time | 4
Not completed — On leave (e.g., parental leave) | 3
Not completed — Non-clinical employee | 1
Not completed — Provider does not see clients | 3
Not completed — Other | 5
Period: Youth Patient Enrollment
Arm/Group | Training Intervention
Started | 125 (Number of GMY identified in partner clinic's electronic health records.)
Completed | 125
Not Completed | 0
Period: Parents of Youth Patient Enrollment
Arm/Group | Training Intervention
Started | 68 (Number of parents of GMY who completed measures related to their youth)
Completed | 68
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Training Intervention: The single-arm intervention study will test an online asynchronous. training intervention.
  The training is a modular online asynchronous training intervention designed to increase mental health providers' use of evidence-based practices with youth patients (ages 12-25). It was developed using community-engaged and human-centered design methods with key stakeholders (youth patients, their parents, mental health providers). In this open trial, the training will be offered to mental health providers at a multisite mental health clinic in the U.S. (referred to as "pilot site" herein).
Arm/Group | Training Intervention
Number analyzed (Participants) | 286
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The overall baseline participant N = 286 is the sum of N = 93 provider, N = 125 youth, and N = 68 parents.
  years
    Providers: number analyzed (Participants) | 93
    Providers | 37 (9)
    Youth Patients: number analyzed (Participants) | 125
    Youth Patients | 16 (3)
    Parents of Youth Patients: number analyzed (Participants) | 68
    Parents of Youth Patients | NA (NA) — Parents did not provide their age
Age, Customized [Count of Participants; unit: Participants] — Population: The overall baseline participant N = 286 is the sum of N = 93 provider, N = 125 youth, and N = 68 parents.
  Participants
    Providers: number analyzed (Participants) | 93
    Providers: >18 | 0
    Providers: 18-65 | 81
    Providers: 65< | 2
    Providers: Not reported | 10
    Youth Patients: number analyzed (Participants) | 125
    Youth Patients: >18 | 51
    Youth Patients: 18-65 | 74
    Youth Patients: 65< | 0
    Youth Patients: Not reported | 0
    Parents of Youth Patients: number analyzed (Participants) | 68
    Parents of Youth Patients: >18 | 0
    Parents of Youth Patients: 18-65 | 0
    Parents of Youth Patients: 65< | 0
    Parents of Youth Patients: Not reported | 68
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The overall baseline participant N = 286 is the sum of N = 93 provider, N = 125 youth, and N = 68 parents.
  Participants
    Providers: number analyzed (Participants) | 93
    Providers: Cisgender Women | 66
    Providers: Cisgender Men | 13
    Providers: Transgender Women | 0
    Providers: Transgender Men | 0
    Providers: Nonbinary/genderqueer | 4
    Providers: Not Reported | 10
    Youth Patients: number analyzed (Participants) | 125
    Youth Patients: Cisgender Women | 0
    Youth Patients: Cisgender Men | 0
    Youth Patients: Transgender Women | 10
    Youth Patients: Transgender Men | 14
    Youth Patients: Nonbinary/genderqueer | 58
    Youth Patients: Not Reported | 43
    Parents of Youth Patients: number analyzed (Participants) | 68
    Parents of Youth Patients: Cisgender Women | 45
    Parents of Youth Patients: Cisgender Men | 18
    Parents of Youth Patients: Transgender Women | 0
    Parents of Youth Patients: Transgender Men | 0
    Parents of Youth Patients: Nonbinary/genderqueer | 0
    Parents of Youth Patients: Not Reported | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall baseline participant N = 286 is the sum of N = 93 provider, N = 125 youth, and N = 68 parents.
  Participants
    Providers: number analyzed (Participants) | 93
    Providers: Hispanic or Latino | 5
    Providers: Not Hispanic or Latino | 78
    Providers: Unknown or Not Reported | 10
    Youth Patients: number analyzed (Participants) | 125
    Youth Patients: Hispanic or Latino | 11
    Youth Patients: Not Hispanic or Latino | 66
    Youth Patients: Unknown or Not Reported | 48
    Parents of Youth Patients: number analyzed (Participants) | 68
    Parents of Youth Patients: Hispanic or Latino | 4
    Parents of Youth Patients: Not Hispanic or Latino | 59
    Parents of Youth Patients: Unknown or Not Reported | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The overall baseline participant N = 286 is the sum of N = 93 provider, N = 125 youth, and N = 68 parents.
  Participants
    Providers: number analyzed (Participants) | 93
    Providers: American Indian or Alaska Native: | 0
    Providers: Asian: | 6
    Providers: Black or African American: | 2
    Providers: Native Hawaiian or Other Pacific Islander: | 0
    Providers: White: | 65
    Providers: More than one race: | 4
    Providers: Other: | 5
    Providers: Unknown: | 11
    Youth Patients: number analyzed (Participants) | 125
    Youth Patients: American Indian or Alaska Native: | 2
    Youth Patients: Asian: | 6
    Youth Patients: Black or African American: | 5
    Youth Patients: Native Hawaiian or Other Pacific Islander: | 0
    Youth Patients: White: | 50
    Youth Patients: More than one race: | 15
    Youth Patients: Other: | 0
    Youth Patients: Unknown: | 47
    Parents of Youth Patients: number analyzed (Participants) | 68
    Parents of Youth Patients: American Indian or Alaska Native: | 0
    Parents of Youth Patients: Asian: | 7
    Parents of Youth Patients: Black or African American: | 1
    Parents of Youth Patients: Native Hawaiian or Other Pacific Islander: | 0
    Parents of Youth Patients: White: | 52
    Parents of Youth Patients: More than one race: | 2
    Parents of Youth Patients: Other: | 0
    Parents of Youth Patients: Unknown: | 6
Region of Enrollment [Number; unit: participants]
  United States | 286

OUTCOME MEASURES:

1. Primary Outcome: Provider Participant Recruitment Rates (Feasibility of Conducting a Larger Trial)
Description: Percent of providers at pilot site who consented to participate in the study relative to number of employed providers at pilot site.
Time Frame: At time of training intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Training Intervention
Number analyzed (Participants) | 109
Participants | 93

2. Primary Outcome: Change in Provider Participant Assessment Completion Rates at Post-training (Feasibility of Conducting a Larger Trial)
Description: Change in the percent of providers who complete pre- and post- assessments of those who consented to participate. These assessment completion rates will also be compared to the 6- and 12-month assessment completion rates.
Time Frame: Pre-training to post-training (up to 4 weeks after the training)
Measure: Count of Participants; unit: Participants
Arm/Group | Training Intervention
Number analyzed (Participants) | 93
Participants | 79

3. Primary Outcome: Change in Provider Participant Assessment Completion Rates at 6-month Followup (Feasibility of Conducting a Larger Trial)
Description: Change in the percent of providers who complete post- and 6-month followup assessments of those who consented to participate. These assessment completion rates will also be compared to the pre-training and 12-month assessment completion rates.
Time Frame: Post-training (up to 4 weeks after the training) to 6-month followup
Measure: Count of Participants; unit: Participants
Arm/Group | Training Intervention
Number analyzed (Participants) | 93
Participants | 47

4. Primary Outcome: Change in Provider Participant Assessment Completion Rates at 12-month Followup (Feasibility of Conducting a Larger Trial)
Description: Change in the percent of providers who complete 6- and 12-month followup assessments of those who consented to participate. These assessment completion rates will also be compared to the pre-training and post-training assessment completion rates.
Time Frame: 6-month followup to 12-month followup
Measure: Count of Participants; unit: Participants
Arm/Group | Training Intervention
Number analyzed (Participants) | 93
Participants | 46

5. Primary Outcome: Change in the Adoption of Practices Learned in the Training Intervention at 12-month Followup
Description: A self-report survey measuring whether, and the extent to which, provider participants used the practices they learned in the training intervention. The survey is currently being developed and will be adapted based on the Pachankis et al. (2022) measure Providers' Familiarity With and Use of LGBTQ-affirmative CBT Skills. The survey will be administered at the 6- and 12 month followups to see the change over time. Scores are calculated using mean scores for values 0-4 with higher numbers indicating more of the use of the practice (i.e., (0) Not at all, (4) Very much)
Time Frame: Baseline, Post-training, 6-month to 12-month followup
Population: Some provider participants did not complete adoption measures at certain time-points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Training Intervention
Number analyzed (Participants) | 93
score on a scale
  Baseline: number analyzed (Participants) | 70
  Baseline | 2.76 (0.73)
  Post-training: number analyzed (Participants) | 70
  Post-training | 3.21 (0.68)
  6-month follow-up: number analyzed (Participants) | 48
  6-month follow-up | 2.86 (0.73)
  12-month follow-up: number analyzed (Participants) | 46
  12-month follow-up | 3.31 (0.51)

6. Primary Outcome: Electronic Monitoring of Training Intervention Completion (Adoption of Training Intervention)
Description: Electronic monitoring of training intervention completion by providers (i.e., whether all modules were completed).
Time Frame: up to the 12-month followup
Measure: Count of Participants; unit: Participants
Arm/Group | Training Intervention
Number analyzed (Participants) | 93
Participants | 78

7. Primary Outcome: Primary Outcome: Electronic Monitoring of Training Intervention Engagement (Adoption of Training Intervention)
Description: Electronic monitoring of training intervention engagement (e.g., days spent completing the training)
Time Frame: up to the 12-month followup
Population: Of the 93 participants who started the training, 78 completed the training. Thus, those 78 providers were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Training Intervention
Number analyzed (Participants) | 78
Days | 18.88 (31.2)

8. Secondary Outcome: Client Behavioral Engagement by Session Participation
Description: Available chart data from clients of providers who completed the intervention will be monitored for their behavioral engagement. Session participation will be measured by electronic health record monitoring of treatment measures completion (e.g., answering all questions and submitting measures related to client treatment, such as the TAQs).
Time Frame: Weekly from pre-intervention to 12 months after training intervention completion
Measure: Count of Participants; unit: Participants
Arm/Group | Training Intervention
Number analyzed (Participants) | 193
Participants
  Youth Patients | 125
  Parents of Youth Patients | 68

9. Secondary Outcome: Client Behavioral Engagement by Session Attendance
Description: Available chart data from clients of providers who completed the intervention will be monitored for their behavioral engagement. Session attendance will be measured as an aspect of behavioral engagement by noting attended and canceled sessions. Outcomes report the total number of GMY participants who attended therapy during the timeframe
Time Frame: Weekly from pre-intervention to 12 months after training intervention completion
Measure: Count of Participants; unit: Participants
Arm/Group | Training Intervention
Number analyzed (Participants) | 125
Participants | 125

10. Secondary Outcome: Therapeutic Alliance Quality Scale (Client Satisfaction & Attitudinal Engagement)
Description: The Therapeutic Alliance Quality Scale (TAQS) is a 5-item questionnaire that asks clients and their caregivers to reflect on their last session with their therapist. Items are rated on a 5-point scale with higher responses corresponding to higher quality alliance (e.g., 1= "Not at all," 2= "Only a little," 3= "Somewhat," 4= "Quite a bit," and 5= "Totally"). The TAQS will be administered to clients aged 12-25 and caregivers. Outcomes report pre-intervention TAQs score (i.e., first instance of participant completing TAQs prior-to intervention) and 12-month follow-up TAQs score.
Time Frame: Weekly from pre-intervention to 12-month follow up
Population: 52 total participants completed the TAQS measure. 3 youth participants completed the measure both at the pre- and 12-month follow-up timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Training Intervention
Number analyzed (Participants) | 52
score on a scale
  Youth Patients, Pre-intervention: number analyzed (Participants) | 27
  Youth Patients, Pre-intervention | 3.72 (.76)
  Youth Patients, 12-month Follow-up: number analyzed (Participants) | 12
  Youth Patients, 12-month Follow-up | 3.95 (1.14)
  Parents of Youth Patients, Pre-Intervention: number analyzed (Participants) | 16
  Parents of Youth Patients, Pre-Intervention | 2.11 (1.17)

11. Secondary Outcome: Service Satisfaction Scale (Client Satisfaction & Attitudinal Engagement)
Description: The Service Satisfaction Scale (SSS) is a 5-item questionnaire that asks clients and their caregivers to reflect on how satisfied they are with the mental health services that they receive. Items are rated on a 4-point scale with higher responses corresponding to higher service satisfaction (e.g., 1= "No, definitely not," 2= "No, not really," 3= "Yes, generally," and 4= "Yes, definitely"). The SSS will be administered to clients aged 12-25 and caregivers. Outcomes report pre-intervention SSS score (i.e., first instance of participant completing SSS prior-to intervention) and 12-month follow-up SSS score.
Time Frame: Every other week from pre-intervention to 12-month follow up
Population: 60 participants total completed the SSS measure. 3 youth participants and 1 caregiver participants completed the measure at both the pre- and 12-month follow-up timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Training Intervention
Number analyzed (Participants) | 60
score on a scale
  Youth Patients, Pre-intervention: number analyzed (Participants) | 27
  Youth Patients, Pre-intervention | 3.25 (0.44)
  Youth Patients, 12-month follow-up: number analyzed (Participants) | 12
  Youth Patients, 12-month follow-up | 3.65 (0.46)
  Parents of Youth Patients, pre-intervention: number analyzed (Participants) | 18
  Parents of Youth Patients, pre-intervention | 3.12 (0.63)
  Parents of Youth Patients, 12-month follow-up: number analyzed (Participants) | 7
  Parents of Youth Patients, 12-month follow-up | 3.96 (0.09)

12. Secondary Outcome: Treatment Outcomes Expectation Scale (Client Satisfaction & Attitudinal Engagement)
Description: The Treatment Outcomes Expectation Scale (TOES) is a 8-item questionnaire that asks clients and their caregivers about their expectations from counseling. Items are rated on a 3-point scale with higher responses corresponding to more expectations (e.g., 1= "I do not expect this," 2= "I am not sure", and 3= "I do expect this"). The TOES will be administered to clients aged 12-25 and caregivers.
Time Frame: Pre-intervention
Population: 47 participants total completed the TOES measure. 23 youth participants and 24 caregiver participants completed the measure at pre-intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Training Intervention
Number analyzed (Participants) | 47
score on a scale
  Youth Patients, Pre-intervention: number analyzed (Participants) | 23
  Youth Patients, Pre-intervention | 2.4 (0.43)
  Parents of Youth Patients, Pre-intervention: number analyzed (Participants) | 24
  Parents of Youth Patients, Pre-intervention | 2.62 (0.28)

13. Secondary Outcome: Treatment Process Expectations Index (Client Satisfaction & Attitudinal Engagement)
Description: The Treatment Process Expectations Index is a 9-item questionnaire that asks clients and their caregivers about their expectations about counseling. Items are rated on a 3-point scale (e.g., 1= "I do not expect this," 2= "I am not sure", and 3= "I do expect this"). There is no right or wrong answer. The reported scores should be interpreted at the item level to identify clinical suggestions for providers based on the clients reported expectations at baseline. The TPEI will be administered to clients aged 12-25 and caregivers.
Time Frame: Pre-intervention
Population: TPEI items are interpreted at the item level and are not scored together; therefore, outcomes report the number of participants who completed the measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Training Intervention
Number analyzed (Participants) | 125
Participants
  Youth Patients, Pre-intervention | 23
  Parents of Youth Patients, Pre-intervention | 24

14. Secondary Outcome: Ohio Functioning Scale (Client Functioning)
Description: The Ohio Functioning Scale is a 20-item questionnaire that asks clients and their caregivers to answer questions regarding how the client's problems may get in the way of everyday activities. Items are rated on a 5-point scale with higher responses corresponding to better ability to do everyday activities (e.g., 0= "Extreme troubles," 1= "Quite a few troubles," 2= "Some troubles", 3= "Ok," and 4= "Doing very well"). A total functioning score ranges from 20-100 and is calculated by summing the ratings for all 20 items. Higher scores are indicative of better functioning. The Ohio Functioning Scale will be administered to clients aged 12-25 and caregivers. Outcomes report pre-intervention Ohio score (i.e., first instance of participant completing Ohio prior-to intervention) and 12-month follow-up Ohio score.
Time Frame: Monthly from pre-intervention to 12-month follow up
Population: 56 participants total completed the OHIO measure. 2 youth participants and 1 caregiver participant completed the measure at both the pre- and 12-month follow-up timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Training Intervention
Number analyzed (Participants) | 56
score on a scale
  Youth Patients, Pre-intervention: number analyzed (Participants) | 27
  Youth Patients, Pre-intervention | 37.3 (11.63)
  Youth Patients, 12-month follow-Up: number analyzed (Participants) | 9
  Youth Patients, 12-month follow-Up | 59.89 (12.57)
  Parent of Youth Patients, Pre-intervention: number analyzed (Participants) | 17
  Parent of Youth Patients, Pre-intervention | 33.88 (16.87)
  Parent of Youth Patients, 12-month follow-up: number analyzed (Participants) | 6
  Parent of Youth Patients, 12-month follow-up | 62.33 (6.59)

15. Secondary Outcome: Symptoms and Functionality Severity Scale (Client Symptomatology & Functioning)
Description: The Symptoms and Functionality Severity Scale which is a 13-item questionnaire that asks clients and their caregivers to reflect on behaviors, thoughts, and feelings that the client had in the last 2 weeks. Items are rated on a 5-point scale with higher responses corresponding to more frequent experiences of negative behaviors, thoughts, and feelings (e.g., 1= "Never," 2= "Hardly Ever," 3= "Sometimes," 4= "Often," and 5= "Very Often"). Scores can range from 33 to 86 for youths, where a high score represents high severity and a low score indicates low severity. Total scores are calculated by adding the rating and then divide the sum by the number of items to calculate the average score.The SFSS will be administered to clients aged 12-25 and caregivers. Outcomes report pre-intervention SFSS score (i.e., first instance of participant completing SFSS prior-to intervention) and 12-month follow-up SFSS score.
Time Frame: Monthly from pre-intervention to 12-month follow up
Population: 67 participants total completed the SFSS measure. 2 youth participants and 3 caregiver participants completed the measure at both the pre- and 12-month follow-up timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Training Intervention
Number analyzed (Participants) | 67
score on a scale
  Youth Patients, Pre-intervention: number analyzed (Participants) | 32
  Youth Patients, Pre-intervention | 52.11 (8.47)
  Youth Patients, 12-month follow-up: number analyzed (Participants) | 9
  Youth Patients, 12-month follow-up | 46 (5.14)
  Parents of Youth Patients, Pre-intervention: number analyzed (Participants) | 25
  Parents of Youth Patients, Pre-intervention | 44.58 (5.89)
  Parents of Youth Patients, 12-month follow-up: number analyzed (Participants) | 6
  Parents of Youth Patients, 12-month follow-up | 38.67 (2.42)

ADVERSE EVENTS:
Time Frame: 2 years, 10 months, and 27 days
Groups:
- Providers: Providers at partner clinic identified as eligible for the study
- Youth Patient: Youth patients identified in partner clinic's electronic health records
- Parents of Youth Patient: Parents of youth patient who completed measures related to their youth
Arm/Group | Providers | Youth Patient | Parents of Youth Patient
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/125 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/125 | 0/68
Other Adverse Events (participants affected / at risk) | 0/109 | 0/125 | 0/68

LIMITATIONS AND CAVEATS:
The primary pilot site changed EHR systems in May 2024, which was near the end of our EHR-data-collection period for this study (18 months; spanning November 2022 to July 2024). Because of this, patients did not complete any surveys in May 2024. We used best statistical practices for handling systematically missing data during data analysis (e.g., multiple imputation). We will also report this missingness in any publication of pilot results involving these data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT05626231/Prot_SAP_ICF_000.pdf